CLINICAL TRIAL: NCT01391728
Title: Active Lifestyle All Your Life-an Intervention Programme for Preventing Fall Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Hans Jonsson/Docent, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20102011
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2011-06

CONDITIONS: Frequency of Accidental Falls; Participation; Self-rated Health; Occupational Gaps

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Active Lifestyle all your Life
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Active Lifestyle all your Life — Intervention After the first data collection the participants are randomised in an intervention and control group. The control group receives the normal treatment that may be given after a radius fracture and may vary from one care unit to another (but there is no preventive programme within the normal activity as far as we know). In groups of 6-8 participants the intervention group starts the programme "Active lifestyle all your life" with group meetings around every other week (10-12 times) and with 2 individual meetings directed at discussing fall risks in the participant's own home environment. After a summer break, Christmas and New Year three follow-up meetings take place, one of which is an individual meeting. The intervention is then terminated, but the participants are encouraged to continue the activity themselves.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of the project is to formulate, implement and evaluate a new type of activity-orientated, evidence-based prevention programme to prevent fall injuries among elderly people. The question examined by the study is whether the intervention programme can:

* significantly reduce accidents and incidents involving falling among the participants,
* influence variables such as satisfaction with life, confidence in one's own ability and a feeling of involvement,
* be shown to be cost effective in terms of the use of resources. The intervention programme - Active lifestyle all your life - is being developed in and for primary care for the cost effective prevention of fall injuries among elderly people using a method that results in continued active life. The aim is to ensure that the elderly person is able to continue living an active life with commitment and involvement, which can in itself prevent fall injuries. This presupposes a knowledge of how to avoid fall injuries and the measures and aids that are available to prevent such injuries. The programme will also provide the participants with a social community in self-supporting groups which, by their own efforts but also with social support, are able to continue some of the activities provided through primary care.

ELIGIBILITY:
Inclusion Criteria:

* 65 or older
* Fall injury in the form of radius fracture or other minor documented fall injury, or one or more fall incidents reported in the last six months (reported to a district nurse in the 75-year discussion)

Exclusion Criteria:

* Cognitive impairments
* Documented psychiatric problems that make participation in organized group activity impossible
* Considerable difficulties in speaking and understanding Swedish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Accidental falls | Two Years (2010-2012)

SECONDARY OUTCOMES:
Participation Self-Rated health Self efficacy | Two Years (2010-2012)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden